CLINICAL TRIAL: NCT04141254
Title: Impact of Early Debriefing and Enhanced Educative Components on Direct Oral Anticoagulant Adherence After Venous Thromboembolism. The DEBRIEF-VTE Study
Brief Title: Impact of Early Debriefing and Enhanced Educative Components on Direct Oral Anticoagulant Adherence After Venous Thromboembolism.
Acronym: DEBRIEF-VTE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 29BRC18.0198
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Venous Thromboembolism
Keywords: Anticoagulant; Direct oral anticoagulant; Debriefing; Recurrent venous thromboembolism; anticoagulant-related bleeding
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: It is a multicenter, randomized trial with blind evaluation, parrallel arm, and using a Zelen randomization process
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Debriefing (Experimental): a standardized follow-up visit at one month associated with "debriefing and enhanced educative component"
  Interventions: Other: Debriefing and educative components
- Without debriefing (Other): a standardized follow-up visit at one month alone (i.e.; without "debriefing and educative component")
  Interventions: Other: Without debriefing and educative components

INTERVENTIONS:
Other: Debriefing and educative components — The patient will receive early debriefing and enhanced educative components added to a standardized visit at one month
  Arms: Debriefing
Other: Without debriefing and educative components — Patient will receive a standardized visit alone (without debriefing and enhanced educative components ) at one month
  Arms: Without debriefing

SUMMARY:
Venous thromboembolism (VTE) is a frequent multifactorial and potential life-threatening disease. Once VTE has been diagnosed, anticoagulation should be started and prolonged for at least three to six months in order to reduce the risk of fatal and non-fatal recurrences and long-term sequelae. The development of direct oral anticoagulants (DOACs) has represented a major advance in patients' care as there is evidence that DOACs are associated with a decreased risk of bleeding without loss in efficacy and as it simplifies treatment modalities for the patients and the physician. However, as DOACs do not require laboratory monitoring, adherence of anticoagulation is difficult to evaluate and traditional programs built on patients receiving VKA may no longer be applicable to patients on DOAC. In order to increase treatment adherence in patients on DOAC for an acute VTE and to improve the quality of life, the impact of specific educational programs on DOACs, taking in account both therapeutic (DOAC) and medical illness (VTE) dimensions needs to be investigated.

In patients with an acute episode of VTE treated for at least 6 months, the main hypothesis is that early debriefing and educative components added to a standardized visit one month after an acute VTE has the potential to improve patient's adherence to APIXABAN therapy at 6 months of follow-up.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a frequent multifactorial and potential life-threatening disease. Once VTE has been diagnosed, anticoagulation should be started and prolonged for at least three to six months in order to reduce the risk of fatal and non-fatal recurrences and long-term sequelae. The development of direct oral anticoagulants (DOACs) has represented a major advance in patients' care as there is evidence that DOACs are associated with a decreased risk of bleeding without loss in efficacy and as it simplifies treatment modalities for the patients and the physician. However, as DOACs do not require laboratory monitoring, adherence of anticoagulation is difficult to evaluate and traditional programs built on patients receiving VKA may no longer be applicable to patients on DOAC. In order to increase treatment adherence in patients on DOAC for an acute VTE and to improve the quality of life, the impact of specific educational programs on DOACs, taking in account both therapeutic (DOAC) and medical illness (VTE) dimensions needs to be investigated.

Design The "DEBRIEF-VTE" trial is a multicenter randomized trial with blind evaluation and using a Zelen randomization process comparing a standardized follow-up visit at one month associated with a "debriefing and enhanced educative components" versus a standardized follow-up visit at one month alone (i.e.; without debriefing process).

All patients meeting the inclusion and none of the exclusion criteria are eligible for randomization. They will be randomized 1:1 to one of two allocated groups:

* Experimental group: a standardized follow-up visit at one month associated with "debriefing and enhanced educative component"
* Control group: a standardized follow-up visit at one month alone (i.e.; without "debriefing and educative component") Randomization will be performed using a two-step methodology described by Zelen et al.
* Stratification by:

  * Center
  * DVT or PE
  * Presence of a major risk factor (either transient or persistent) or not (unprovoked VTE) At visit 1 (inclusion, 0-7 days): Inclusion of patients using the first written informed consent to accept a standard follow-up (visit at 1 month and 6 months) without mentioning randomization at one month performed in order to allocate patients to have, or to not have, debriefing and enhanced educative components. Study medication will be administered with complete explanation about doses and a classical therapeutic information regarding DOAC and clinical signs of recurrent VTE and bleeding (one treatment box with 400 pills of apixaban at 5 mg for the first 6 months of therapy) will be performed.

Visit 2 (30 days):

* Before the visit 2, review of all the inclusion and exclusion criteria and compute creatinine clearance using Cockcroft-Gault method ; if all eligibility criteria are satisfied, randomization of the patient;
* After randomization, during the visit 2:

  * For patients allocated to the experimental group: signature of the second written informed consent describing the debriefing and enhanced educative components and objective on quality of life
  * For patients allocated to the control group: no second written informed consent is required

Visit 3/ET (180 days):

- Evaluate quality of life (PembQOL if PE, VEINES-Qol if DVT, EQ-5D for all patients), residual symptoms (mMRC and MDP scale if PE, Villalta if DVT) depression (HAD), recurrent VTE, bleeding, hospitalizations, death

The primary objective is to demonstrate that, in patients with an acute episode of VTE treated for at least 6 months, early debriefing and enhanced educative components added to a standardized visit one month after an acute VTE is associated with an increased adherence to apixaban therapy at 6 months than after a standardized visit alone at one month (adherence measured by the MEMSCap™ Medication Event Monitoring System Cap (WestRock, USA & Switzerland). In patients with an acute episode of VTE treated for at least 6 months, the main hypothesis is that early debriefing and educative components added to a standardized visit one month after an acute VTE has the potential to improve patient's adherence to APIXABAN therapy at 6 months of follow-up.

Secondary objectives are to evaluate the impact of early debriefing and enhanced educative components added to a standardized visit one month after an acute VTE on the following at 6 months of treatment : quality of life (EQ-5D for all, PembQOL if PE, VEINES-Qol if DVT), residual symptoms (MMRC and multidimensional dyspnea profile(MDP) scales if PE, Villalta if DVT), depression (HAD), recurrent VTE, bleeding,hospitalizations and death.

150 patients will be included Duration of the inclusion period: 18 months Duration of participation for each patient: 6 months Total duration of the study: 24 months

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old, the upper limit of which will be left to the discretion of the investigator according to the risk benefit balance
* Patients with indications for a minimum of 6 months of anticoagulation after an acute documented VTE that was diagnosed 7 days ago or less (i.e.; symptomatic PE or proximal or distal DVT)
* Social security affiliation.
* Patient who signed inform consent form

Exclusion Criteria:

* Known allergy to apixaban, allergy to any of the excipients
* Unable or refusal to give informed consent
* Indication for anticoagulation other than DVT or PE (e.g.; atrial fibrillation, mechanic valves…)
* Treatment with investigational drug in the past 1 month
* Chronic liver disease or chronic hepatitis
* Renal insufficiency with creatinine <30 ml / min on Cockcroft and Gault formula
* Known antiphospholipid syndrome
* Dual anti-platelet therapy or aspirin at dosage >100 mg per day
* Concomitant use of a strong inhibitor of cytochrome P450 3A4 (CYP3A4) (e.g., a protease inhibitor for human immunodeficiency virus infection or azole-antimycotics agents ketoconazole, itraconazole, voriconazole, posaconazole) or a CYP3A4 inducer (e.g., rifampin, carbamazepine, or phenytoin),
* Active cancer of less than 6 months
* Active pregnancy or expected pregnancy in the next 6 months
* Planned surgery in the next 6 months
* No effective contraception in women of childbearing age
* Life expectancy <6 months
* Patient with active clinically significant bleeding
* Patient with lesion or condition if considered a significant risk factor for major bleeding
* Patient with concomitant treatment with any other anticoagulant agent
* Patient with concomitant treatment as: P-gp inhibitors: ciclosporin, dronedarone, quinidine, verapamil, protease inhibitors (e.g.: ritonavir, nelfinavir, indinavir, saquinavir), macrolides (e.g.; erythromycin, clarithromycine), azole antifungals (e.g.; ketoconazole, itraconazole, voriconazole, posaconazole).
* Patient with concomitant treatment as non steroidal antiinflammatory drugs
* Patient with low body weight (< 60kg).
* Patients with breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence mesured by Medication Event Monitoring System Cap | at 6 months
  Adherence to apixaban therapy at 6 months after an acute episode of VTE measured by the MEMSCap™ will be evaluated.
  The main criteria for adherence measurement will be the number of days where patients took adequately apixaban divided by the number of expected days of prescription. An additional evaluation will be the number of taken pills divided by the expected taken pills.

SECONDARY OUTCOMES:
Treatment adherence mesured by Medication Event Monitoring System Cap | at 1 month and 3 months
  Adherence to apixaban therapy at 1 month and 3 months after an acute episode of VTE measured by the MEMSCap™ will be evaluated.
  The main criteria for adherence measurement will be the number of days where patients took adequately apixaban divided by the number of expected days of prescription. An additional evaluation will be the number of taken pills divided by the expected taken pills.
Quality of life after an acute VTE | At 6 months
  Quality of life of patients with VTE will be evaluated by the EQ-5D questionnaire
Quality of life after an acute VTE | At 6 months
  Quality of life of patients with VTE will be evaluated by the HAD scale
Recurrent VTE (Symptomatic recurrent pulmonary embolism and Symptomatic recurrent deep-vein thrombosis) diagnosed on the basis of a clinical suspicion | during a study treatment period of 6 months
  Adjudicated symptomatic objectively confirmed recurrent VTE (non fatal or fatal VTE) during the study treatment period
Major and clinically relevant non major bleeding | during a study treatment period of 6 months
  Adjudicated major bleeding (as defined by the criteria of the International Society of Thrombosis and Haemostasis) or clinically relevant non major bleeding during the study treatment period
Mortality | during a study treatment period of 6 months
  Mortality due to VTE, bleeding or other cause than recurrent VTE or major or clinically relevant non major bleeding during the study treatment period will be adjudicated
Hospitalisation for an acute medical illness during treatment period will be evaluated by questioning the patient | during a study treatment period of 6 months
  Hospitalization for an acute medical illness during treatement period will be evaluated by questioning the patient

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Angers, Angers
  - HIA Brest, Brest
  - CHRU de Brest, Brest
  - CHU de Clermont Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - APHP Hôpital Louis Mourier, Colombes
  - CHU de Grenoble - Hôpital Nord Michallon, Grenoble
  - HEGP, Paris
  - CHU de Rennes - Hôpital Sud, Rennes
  - CHU de Saint Etienne - Hôpital Nord, Saint-Etienne
  - CHU de Toulouse - Hôpital de Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No